CLINICAL TRIAL: NCT06044428
Title: Steadysense -Early Detection of Postoperative Infections Through Continuous Temperature Measurement
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Ek-Nr.: 35-251 ex 22/23
Record Dates: First submitted 2023-08-28; First posted 2023-09-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Body Temperature; Postoperative Infection; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Steadytemp® — Steadytemp® is a clinical thermometer intended to continuously measure axillary temperature and to display relative changes in axillary temperature to the user. The system consists of a sensor patch and a smartphone application, the body temperature measured by the sensor is transmitted via Near-Field-Communication (NFC) and subsequently displayed in the App.

SUMMARY:
The goal of this observational study is to review whether postoperative infections can be detected earlier by a continuous measurement of body temperature of patients compared to single daily measurements. Within 25 weeks 100 patients, which underwent visceral surgery less than 48h ago, will be included. A patch (Steadytemp ®) will be attached to participants, continuously measuring the body temperature. In addition infection parameters and medication of the participants will be documented.

ELIGIBILITY:
Inclusion Criteria:

* participant is willing and able to give informed consent for participation in the study
* age 18 years and above
* visceral surgery procedure within the last two days
* inpatient stay on the ICIÜ (Interdisciplinary surgical intensive care unit) or normal ward

Exclusion Criteria:

* allergy to the ingredients of skin patches
* major psychiatric diseases including history of drug or alcohol abuse
* chronic inflammatory disease in the medical history
* predicted inpatient stay is less than 5 days
* operational wound is too close to the patch adhesive site
* the skin at the intended adhesive site of the patch is not intact
* BMI > 33

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be inpatients at the Medical University of Graz, where the need to have a visceral surgery.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Temperature curve (body temperature in °C) | min. 5 days and max. 21 days
  temperature curve of the Steadytemp® Patch and single routine measurements (infrared)
wound infection or pneumonia | min. 5 days and max. 21 days
  Number of patients diagnosed with wound infection or pneumonia

SECONDARY OUTCOMES:
Inflammation parameter in the blood: PCT (Procalcitonin) | min. 5 days and max. 21 days
  PCT (Procalcitonin) level
Inflammation parameter in the blood: CRP (c-reactive protein) | min. 5 days and max. 21 days
  CRP (c-reactive protein) level
Inflammation parameter in the blood: Leukocytes | min. 5 days and max. 21 days
  Leukocytes count
Use of medication | min. 5 days and max. 21 days
  Use of medication like antibiotics, antiphlogistics, antipyretics

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Philipp Stiegler, Assoc. Prof., Principal Investigator — Medical University Graz, Department of Surgery, Division of general, visceral and transplant surgery
Locations (1):
- Medical University of Graz, Graz, Austria